CLINICAL TRIAL: NCT01878097
Title: Green Dot Across the Bluegrass: Evaluation of a Primary Prevention Intervention
Brief Title: Evaluation of Green Dot a Primary Prevention Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Ann Coker, Professor and Endowed Chair, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5U01CE001675 (NIH)
Record Dates: First submitted 2013-03-29; First posted 2013-06-14 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Sex Offenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Green Dot Bystander Training (Experimental): Green Dot intervention
  Interventions: Behavioral: Green Dot Bystander Intevention
- Control (Active Comparator): Awareness Eduation
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Green Dot Bystander Intevention — Intervention allocated at the school level
  Arms: Green Dot Bystander Training
Behavioral: Control — Awareness Education
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the statewide application of Green Dot among high schools students. We hypothesize that students in high schools with Green Dot will over time report lower rates of sexual violence (SV) compared with students in comparable high schools randomized not to have Green Dot. This reduction in sexual violence will be mediated through a reduction in social norms supporting sexual violence (measured with violence acceptance scales) and an increase in bystander behaviors.

DETAILED DESCRIPTION:
"Green Dot" is a bystander intervention program that empowers students to actively question peer support for sexual violence (SV) and become change agents who play a significant role in preventing sexual violence. The purpose of this study is to evaluate the statewide application of Green Dot among high schools students. We hypothesize that students in high schools with Green Dot will over time report lower rates of SV compared with students in comparable high schools randomized not to have Green Dot. A high school based controlled intervention trial is being used to test the efficacy of Green Dot. Both panel and cohort survey methods will be used to provide baseline and prospective data on student's attitudes supporting SV, bystander behaviors and violence victimization and perpetration. In 13 Kentucky regions, 2 demographically comparable high schools were recruited to participate in Green Dot intervention either as the intervention or control site. Schools were randomly assigned to the intervention. Study Population includes all students in participating high schools invited to complete anonymous panel surveys beginning spring 2010 through 2014. This state-wide, population-based, multi-site controlled intervention trial provides an empirical test of a promising intervention, which, if proven effective, could result in the primary prevention of SV and a reduction in the health and academic consequences of SV.

ELIGIBILITY:
Inclusion Criteria:

Only high school students attending the intervention or comparison high schools will be eligible. Two groups will be recruited: those receiving bystanding training and those not receiving such training who may or may not be in the social network of those receiving bystanding training.

Exclusion Criteria:

All other high school students in Kentucky

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 89707 (Actual)
Dates: Start 2009-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann L. Coker, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- [Result] Coker AL, Bush HM, Cook-Craig PG, DeGue SA, Clear ER, Brancato CJ, Fisher BS, Recktenwald EA. RCT Testing Bystander Effectiveness to Reduce Violence. Am J Prev Med. 2017 May;52(5):566-578. doi: 10.1016/j.amepre.2017.01.020. Epub 2017 Mar 6. PMID 28279546
- [Result] Coker AL, Bush HM, Brancato CJ, Clear ER, Recktenwald EA. Bystander Program Effectiveness to Reduce Violence Acceptance: RCT in High Schools. J Fam Violence. 2019;34(3):153-164. doi: 10.1007/s10896-018-9961-8. Epub 2018 Apr 2. PMID 30956390
- [Derived] Mennicke AM, Bush HM, Brancato CJ, Coker AL. Bystander Program to Reduce Sexual Violence by Witnessing Parental Intimate Partner Violence Status. Am J Prev Med. 2022 Aug;63(2):262-272. doi: 10.1016/j.amepre.2021.12.022. Epub 2022 Mar 9. PMID 35279345

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 89,707 students completed surveys. However, due to anonymous response, it is not possible to know the number of unique students who completed surveys within the study period. Two schools within each of the 13 regions were selected by the Rape Crisis Centers for simple randomization to each condition in this cluster RCT (n=26).
Pre-assignment Details: 46 demographically similar public high schools were identified as willing participate in the trial. Two schools were excluded by researchers because these were too small (<100 per grade). Among the remaining 36 schools, two schools within each of the 13 regions were selected and randomized (n=26).
Units Other Than Participants: High schools
Groups:
- Green Dot Bystander Training: 13 receiving Green Dot intervention
  Green Dot Bystander Intevention: Intervention allocated at the school level
- Control: 13 high school receiving no bystander training (no intervention)
Period: Baseline
Arm/Group | Green Dot Bystander Training | Control
Started | 10725; 13 High schools (number of students in 13 intervention schools completing anonymous surveys with non missing data) | 10081; 13 High schools (number of students in 13 control schools completing anonymous surveys with non missing data)
Completed (Anonymous surveys; sum of all completed surveys.) | 8228; 13 High schools (Anonymous surveys so only last year data provided as annual completed.) | 8281; 13 High schools (Anonymous surveys; sum of all completed surveys.)
Not Completed | 2497; 0 High schools | 1800; 0 High schools
Not completed — Surveys not fully completed | 2497 | 1800
Period: Implementation Year 1
Arm/Group | Green Dot Bystander Training | Control
Started | 11742; 13 High schools | 9866; 12 High schools
Completed | 8540; 13 High schools | 7317; 12 High schools
Not Completed | 3202; 0 High schools | 2549; 0 High schools
Not completed — Surveys not fully completed | 3202 | 2549
Period: Implementation Year 2
Arm/Group | Green Dot Bystander Training | Control
Started | 11567; 13 High schools | 9611; 12 High schools
Completed | 8286; 13 High schools | 6770; 12 High schools
Not Completed | 3281; 0 High schools | 2841; 0 High schools
Not completed — Surveys not fully completed | 3281 | 2841
Period: Implementation Year 3
Arm/Group | Green Dot Bystander Training | Control
Started | 10540; 13 High schools | 9750; 12 High schools
Completed | 7046; 13 High schools | 6770; 12 High schools
Not Completed | 3494; 0 High schools | 2980; 0 High schools
Not completed — Surveys not fully completed | 3494 | 2980
Period: Implementation Year 4
Arm/Group | Green Dot Bystander Training | Control
Started | 10585; 12 High schools | 9614; 12 High schools
Completed | 6981; 12 High schools | 6607; 12 High schools
Not Completed | 3604; 0 High schools | 3007; 0 High schools
Not completed — Surveys not fully completed | 3604 | 3007

BASELINE CHARACTERISTICS:
Population: Surveys were anonymous. The number of participants analyzed represents the number of analyzable surveys within each group.
Units Other Than Participants: Schools
Groups:
- Green Dot Bystander Training: 26 high schools: 13 receiving Green Dot intervention and 13 no intervention
  Green Dot Bystander Intevention: Intervention allocated at the school level
- Total: Total of all reporting groups
Arm/Group | Green Dot Bystander Training | Control Training | Total
Number analyzed (Participants) | 30853 | 27516 | 58369
Number analyzed (Schools) | 13 | 13 | 26
Age, Customized [Mean (Standard Deviation); unit: Percentage of Participants per School]
  Year in School: First Year | 31.1 (5.54) | 30.37 (3.3) | 30.69 (4.48)
  Year in School: Sophomore | 27.99 (3.95) | 26.72 (3.69) | 27.35 (3.8)
  Year in School: Junior | 25.2 (5.95) | 26.37 (4.52) | 25.78 (5.21)
  Year in School: Senior | 15.54 (9.94) | 16.45 (7.96) | 16 (8.83)
Sex/Gender, Customized [Mean (Standard Deviation); unit: Percentage of Participants per School]
  Female | 54.56 (3.2) | 54.11 (2.98) | 54.33 (3.04)
  Male | 45.44 (3.2) | 45.89 (2.98) | 45.67 (3.04)
Race/Ethnicity, Customized [Mean (Standard Deviation); unit: Percentage of Participants per School]
  American Indian or Alaska Native | 1.08 (0.56) | 1.13 (0.27) | 1.11 (0.43)
  Asian | 1.44 (1.59) | 1.2 (1.08) | 1.32 (1.33)
  Black or African American | 8.03 (10.77) | 6.47 (8.65) | 7.25 (9.6)
  Hispanic or Latino/Latina | 3.16 (2.99) | 1.31 (0.92) | 2.23 (2.37)
  White | 82.51 (17.06) | 87.22 (11.93) | 84.86 (14.62)
  Other | 3.78 (3.28) | 2.67 (2.21) | 3.23 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Sexual Assault Events Used (Perpetrated) Per School.
Description: Students self report of sexual assault perpetration averaged at the school level and adjusted for baseline and number of students. Adjustments were made by including baseline measure and number of students as a covariate in the model. Data will be collected at baseline and annually for 4 years.
Time Frame: up to 5 years follow up from baseline intervention
Population: Anonymous survey data collected over 5 years and sorted by intervention. To complete ITT analysis, schools that dropped out were included in analysis using imputed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of events per school
Units Other Than Participants: Schools
Groups:
- Green Dot Bystander Training: Phase one and two.
- Control: No bystander intervention
Arm/Group | Green Dot Bystander Training | Control
Number analyzed (Participants) | 30853 | 27516
Number analyzed (Schools) | 13 | 13
Number of events per school
  Year 1: number analyzed (Participants) | 8540 | 7317
  Year 1 | 518 [430 to 605] | 420 [353 to 486]
  Year 2: number analyzed (Participants) | 8286 | 6822
  Year 2 | 485 [406 to 563] | 472 [353 to 552]
  Year 3: number analyzed (Participants) | 7046 | 6770
  Year 3 | 292 [218 to 365] | 459 [392 to 526]
  Year 4: number analyzed (Participants) | 6981 | 6607
  Year 4 | 308 [224 to 392] | 370 [316 to 424]
Statistical Analysis 1: Comparison: Green Dot Bystander Training vs Control; Test type: Superiority; p = 0.0003, Mixed Models Analysis; F-stat = 7.12

2. Primary Outcome: Average Number of Sexual Assaults Experienced (Victimization) Events Per School.
Description: Students self report of sexual assault victimization averaged at the school level and adjusted for baseline and number of students. Adjustments made by including baseline measure and number of students as covariates in models. Data will be collected at baseline and annually for 4 years.
Time Frame: Data will be collected at baseline and annually for 4 years.
Population: anonymous survey data collected over 5 years and sorted by intervention. To keep ITT analysis, all schools were included and data were imputed for schools that dropped out.
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of events per school
Units Other Than Participants: Schools
Arm/Group | Green Dot Bystander Training | Control
Number analyzed (Participants) | 30853 | 27516
Number analyzed (Schools) | 13 | 13
Number of events per school
  Year 1: number analyzed (Participants) | 8540 | 7317
  Year 1 | 300 [234 to 367] | 211 [160 to 262]
  Year 2: number analyzed (Participants) | 8286 | 6822
  Year 2 | 292 [227 to 357] | 269 [218 to 320]
  Year 3: number analyzed (Participants) | 7046 | 6770
  Year 3 | 161 [100 to 223] | 281 [215 to 348]
  Year 4: number analyzed (Participants) | 6981 | 6607
  Year 4 | 157 [100 to 214] | 245 [193 to 297]
Statistical Analysis 1: Comparison: Green Dot Bystander Training vs Control; Test type: Superiority; p = 0.0003, Mixed Models Analysis; F-stat = 7.18

3. Other Pre Specified Outcome: Change in Violence Acceptance
Description: Illinois Rape Myth Acceptance Scale measure students' beliefs about rape which may indicate social norms supporting sexual violence. The scale consists of 22 questions scored 1 -5. Were 1 is "strongly agree" and 5 is "strongly disagree". The higher the cumulative score, the more likely the participant is to accept rape myths.
  5-item Acceptance of General Dating Violence Scale was used to measure norms supporting dating violence. Scores will range from 1-6, were the higher the score the more likely the participant was to reject dating violence as normal.
Time Frame: Data will be collected at baseline and annually for 4 years.
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Increase in Bystanding Behaviors
Description: 7 item survey measuring self-reports of students actively engaging their peers in behaviors that may prevent violence.
  Response options: 0 times, 1-2 times, 3-5 times, 6-9 times, 10 or more times, didn't see or hear someone doing this
  Above items repeated to measure student observing others doing these behaviors. Data will be presented as the total number of interventions were the bigger the number the more likely the bystander was to intervene on behalf of the victim.
Time Frame: Data will be collected at baseline and annually for 4 years.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: No adverse events were monitored in this study
Description: No adverse events were monitored in this study
Groups:
- GreenDot: Experimental: GreenDot Bystander Training "GreenDot" is a bystander intervention program that empowers students to actively question peer support for sexual violence (SV) and become change agents who play a significant role in preventing sexual violence.
- Control: In 13 Kentucky region , 2 demographically comparable high schools were recruited to participate in GreenDot intervention as either the intervention or control site. Schools were randomly assigned to the intervention. Control schools received no additional programming on their campus.
Arm/Group | GreenDot | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Individuals were not tracked over time as surveys were anonymous. Thus, we cannot extrapolate data to make individual conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No